CLINICAL TRIAL: NCT04557085
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Cenobamate Adjunctive Therapy in Subjects With Partial Onset Seizures, With Optional Open-Label Extension
Brief Title: Randomized, Double-blind Study to Evaluate Efficacy and Safety of Cenobamate Adjunctive Therapy in POS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YKP3089C035
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Partial Seizure; Focal Seizure
MeSH Terms: conditions — Seizures | interventions — Cenobamate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Cenobamate 100 mg/day (Experimental): Cenobamate 100 mg/day
  Interventions: Drug: Cenobamate
- Cenobamate 200 mg/day (Experimental): Cenobamate 200 mg/day
  Interventions: Drug: Cenobamate
- Cenobamate 400 mg/day (Experimental): Cenobamate 400 mg/day
  Interventions: Drug: Cenobamate

INTERVENTIONS:
Drug: Cenobamate — Cenobamate tablets
  Arms: Cenobamate 100 mg/day; Cenobamate 200 mg/day; Cenobamate 400 mg/day
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, adjunctive therapy study in subjects with POS, with optional OLE. The study consists of 4 periods as follows: An 8-week of Screening/Baseline Period, 24-week of Double-blind Treatment Period (including a 18-week Titration Phase and 6-week Maintenance Phase), 52-week of Open-label Extension (OLE) Period (applicable for subjects who participate in the OLE) and up to 5-week of End of Study (EOS) Follow-up Period.

The purpose of this study is to evaluate the efficacy and safety of 100, 200 and 400 mg/day of cenobamate as adjunctive therapy compared with placebo in subjects with partial onset seizures (POS).

The study will also evaluate the long-term safety and tolerability of cenobamate adjunctive therapy in subjects with POS who have completed the double-blind treatment period.

DETAILED DESCRIPTION:
Subjects will undergo an 8-week Screening/Baseline Period to assess seizure frequency. Subjects with a high enough number of seizures will be randomized in a 1:1:1:1 ratio to receive placebo or cenobamate 100, 200, or 400 mg given once per day in the morning. Subjects will first enter the 18-week Titration Phase, during which the initial dose will be 12.5 mg/day or placebo. The dose of cenobamate will be increased in a double-blind fashion from 12.5 mg/day to 25 mg/day and 50 mg/day (or matching placebo) at 2-week intervals and then will be titrated by 50 mg/day (or matching placebo) every 2 weeks. After 18-week up-titration, subjects will enter the Maintenance Phase. During the Maintenance Phase, subjects are recommended to maintain their dose for 6 weeks. Subjects who have completed the Double-blind Treatment Period and who choose to participate in this OLE will enter an 18-week Double-blind Conversion Phase before starting the 34-week Open-label Maintenance Phase. Subjects who do not enroll into the OLE will enter a 5-week FU period.

The primary objective of this study is to evaluate the efficacy of cenobamate as adjunctive therapy compared with placebo in subjects with POS. The secondary objectives of this study are: To evaluate the safety and tolerability of cenobamate in subjects with POS, to evaluate the effect of cenobamate in POS and in specified seizure types, and to assess blood plasma exposure of cenobamate in subjects with POS.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following criteria to be enrolled in the study:

1. Male or female subject and age 18 to 70 years inclusive at the time of signing the informed consent
2. Weight at least 35 kg
3. Written informed consent signed by the subject prior to entering the study in accordance with the ICH GCP guidelines. For subjects who lack the capacity, consent will be obtained from the parent/legal guardian. For all underaged subjects according to the specific laws of the country, both the written consent of the subject and the consent of the parent/legal guardian will be obtained.
4. A diagnosis of partial onset seizures according to the International League Against Epilepsy's Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history and an electroencephalogram (EEG).
5. EEG performed within 5 years prior to Visit 1 that is consistent with localization related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (i.e., clinical history). For chronic patients for which the current diagnosis is not very clear, additional EEG results older than 5 years but within 10 years may be used for final confirmation of epilepsy diagnosis.
6. Need additional antiepileptic drug (AED) treatment despite having been treated with at least one AED for the last 2 years.
7. During the 8-week Screening/Baseline Period, subjects must have at least 8 partial seizures including only simple partial seizures with motor component, complex partial seizures, or secondarily generalized seizures without a seizure-free interval of greater than 25 days any time during the 8-week period. Subjects must have at least 3 of these partial seizures during each of the two consecutive 4-week segments of the Screening/Baseline Periods, respectively.
8. Currently on stable antiepileptic treatment regimen:

   1. Subject must have been receiving stable doses of 1 to 3 AEDs for at least 4 weeks prior to Visit 1 to be continued unchanged throughout the Double-blind Treatment Period.
   2. Vagal nerve stimulator (VNS) or deep brain stimulator (DBS) will not be counted as an AED; however, the parameters must remain stable for at least 4 weeks prior to Visit 1 and during the study. VNS or DBS must have been implanted at least 5 months prior to Visit 1.
   3. The daily use of benzodiazepines (except for diazepam) for epilepsy, or for anxiety or sleep disorder, will be counted as 1 AED and must be continued unchanged throughout the study. Therefore, only a maximum of 2 additional approved AEDs will be allowed.
   4. Subjects receiving felbamate as a concomitant AED must meet the following criteria:

   i. Two-year history of felbamate use and a history of a fixed dosing regimen for a minimum of 60 days prior to Visit 1 ii. No prior or known history of hepatotoxicity or hematologic disorder due to felbamate
9. Computed tomography (CT) or magnetic resonance imaging (MRI) scan performed within the past 5 years that ruled out a progressive cause of epilepsy. If brain imaging has not been performed within the past 5 years, a CT scan must be performed prior to randomization. For chronic patients for which the current diagnosis is not very clear, additional CT or MRI results older than 5 years but within 10 years may be used for final confirmation of epilepsy diagnosis.
10. Ability to reach subject by telephone
11. Use of an acceptable form of birth control by female subjects of childbearing potential
12. Subject taking a ketogenic diet will be allowed as long as the diet has been stable for at least 3 months prior to Visit 1 and will remain stable for the duration of the study.

Exclusion Criteria:

1. Female subjects who are pregnant (or planning to become pregnant during the study), lactating or breast-feeding
2. History of non-epileptic or psychogenic seizures
3. Presence of only non-motor simple partial seizures or primary generalized epilepsies
4. History of seizure clusters (episodes lasting less than 30 minutes in which multiple seizures occur with such frequency that the initiation and completion of each individual seizure cannot be distinguished) within 6 months prior to Visit 1
5. Presence or previous history of Lennox-Gastaut syndrome
6. Scheduled epilepsy surgery within 8 months of Visit 1
7. Evidence of any clinically significant laboratory abnormalities or disease (e.g., psychiatric, behavioral problems, cardiac, respiratory, gastrointestinal, hepatic [liver transaminases, ALT or AST, more than twice the upper limit of normal (ULN) or total or direct bilirubin not within normal limits], or renal disease) that, in the opinion of the Investigator, could affect subject's safety or conduct of the study.
8. Any clinically significant active central nervous system (CNS) infection, demyelinating disease, degenerative neurologic disease, or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results
9. Presence of psychotic disorders and/or unstable recurrent affective disorders evident by use of antipsychotics; presence or recent history (within 6 months) of major depressive episode
10. Use of intermittent rescue benzodiazepines more than once per month (1 to 2 doses in a 24-hour period is considered as 1 rescue) in the 1-month period prior to Visit 1
11. Current or recent use (within 30 days prior to Visit 1) of any of the following medications: diazepam/phenytoin/phenobarbital (or metabolites of these drugs), clopidogrel, fluvoxamine, amitriptyline, clomipramine, bupropion, methadone, ifosfamide, cyclophosphamide, efavirenz, natural progesterone, or traditional Chinese/herbal medicines indicated for neurological system
12. Current or recent (within 5 months prior to Visit 1) use of vigabatrin or ezogabine. Subjects with a prior history of treatment with vigabatrin must have documentation showing no evidence of a vigabatrin associated clinically significant abnormality in a visual perimetry test. Subjects with a prior history of treatment with ezogabine should have no evidence of retinal abnormalities with funduscopic features similar to those seen in retinal pigment dystrophies.
13. Previous exposure to cenobamate
14. Participation in any other trials involving an investigational product or device within 30 days prior to Visit 1
15. History of alcoholism, drug abuse, or drug addiction within the past 2 years prior to Visit 1 as assessed by the Investigator
16. History of status epilepticus within 3 months of Visit 1
17. History of any serious drug-induced hypersensitivity reaction (including but not limited to Stevens-Johnson syndrome, toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms [DRESS]) or any drug-related rash requiring hospitalization
18. History of AED-associated rash that involved conjunctiva or mucosae
19. History of any drug-related hypersensitivity reaction that required discontinuation of the medication
20. Presence of Familial short QT syndrome or relevant replicated QTc interval (QTcF less than 340 msec or greater than 450 msec in males and greater than 470 msec in females) on electrocardiogram (ECG)
21. Absolute neutrophil count less than 1,500/μL
22. Platelet counts lower than 80,000/μL in subjects treated with VPA
23. Creatinine clearance less than 60 mL/min, as calculated by Cockcroft-Gault equation
24. History of positive test results for HBsAg, HCV-Ab, and HIV-Ab
25. More than 1 lifetime suicide attempt
26. A "YES" answer to Question 1 or 2 of the C-SSRS (Baseline/Screening version) Suicidal Ideation section in the past 6 months or a "YES" answer to any of the Suicidal Behavior Questions in the past 2 years
27. Subject is a staff member or immediate family member of study staff.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in seizure frequency (seizure rate per 28-day interval) of all simple partial motor, complex partial, or secondarily generalized seizures during the Maintenance Phase. | per 28 days during 6 week maintenance phase

CONTACTS AND LOCATIONS:
Locations (3):
- Site 3, Shanghai, China
- Site 2, Tokyo, Japan
- Site 1, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu X, Chen L, Choe E, Heo K, Hong SB, Iida K, Jeon YH, Jung J, Kamin M, Kawai K, Kim JH, Kim MW, Lee SK, Misra SN, Park J, Rosenfeld WE, Wang T, Yamamoto T, Yu P, Ferrari L. Efficacy of adjunctive cenobamate by focal seizure subtypes: a randomized, double-blind, placebo-controlled, multicenter study in a multinational Asian population. Seizure. 2025 Dec;133:43-51. doi: 10.1016/j.seizure.2025.09.021. Epub 2025 Sep 29. PMID 41101116